CLINICAL TRIAL: NCT06632652
Title: Establish Telenursing System by Providing Health Education and Lifestyle Modification Among Diabetic Patients in Bangladesh
Brief Title: Telenursing System by Providing Health Education and Lifestyle Modification Among Diabetic Patients in Bangladesh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Grameen Caledonian College of Nursing (Unknown)
Responsible Party: Principal Investigator, KATM Ehsanul Huq, Principal Investigator, Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BMRC/NREC/2022-2025/336
Record Dates: First submitted 2024-09-20; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus
Keywords: telenursing; health education; lifestyle modification; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Health Education

STUDY DESIGN:
Intervention Model Description: A quasi-experimental pre- and post-intervention design will be implemented. Investigators will enroll the participants and collect baseline data and then investigators will educate participants, and after 6 months investigators will evaluate participants and compare the baseline (pretest) and endline (posttest) data of individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre- and post-intervention design (Experimental): After enrollment patients receive 'Health Education'. Then patients receive weekly follow up monitoring over phone call for 3 months. After 3 months, patients are requested to visit the Primary Health Care Center (PHC) for follow-up by physician and lab test. From 4-6 months, they receive bi-weekly follow up over phone call and at the end of 6 month, group evaluation for 1 hour and endline data will be collected by the nurses at the PHC.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — Provide 'Health Education' for acquisition of self-management skills, acquiring knowledge of both the disease and self-care. By making self-supported decisions, the patients are able to manage their diet, exercise and medication.
  Patients will start implementing diabetes management right after the group education. Each patient will develop monthly goal settings (behavior change plan) related to their diabetes management, daily practice them, and record the results every day on the self-monitoring notebook. The nurses call each patient on the scheduled day, ask/evaluate his/her behavior changes and monitored data, then make "step-up goals" for the next month. In addition, based on his/her knowledge and practice level, the nurses provide education using the education booklet. Patients and the nurses repeat these activities during 6 months.

SUMMARY:
The global burden of chronic diseases is increasing and becoming a public health issue throughout the world. The use of telenursing is increasing significantly during and after the COVID-19 pandemic to treat and prevent chronic diseases. Study objectives: The objective of this study is to apply the self-management telenursing program and telenursing system developed by the researchers to Bangladesh and to evaluate its feasibility and efficacy (improved diabetes control in participants). Method: This is a pilot, quasi-experimental pre- and post-intervention study. Diabetes patients who will attend the Grameen Primary Health Care Centers (PHCs) in Bangladesh will be enrolled. Investigators include patients who have been diagnosed with type 2 diabetes, both sexes, age above 18-75 years old, all types of treatment, and willing to participate / give consent. Investigators exclude patients who have been diagnosed as gestational diabetes, diabetes as a secondary cause, complication of CKD stage 5, HbA1c is less than 7.0% for past 1 year with CKD stage 1 or 2, no complications or complications with good control, having enough knowledge (had education before) and implemented good practice regarding diabetes management assessed by the research nurses, and disabled persons who need other person's support for daily living. The sample size was calculated and found 70. Patients who meet the eligibility criteria will be introduced by physicians at the PHCs, and the nurses will contact the patients at the PHC. Written informed consent (ICFs) will be obtained from all the participants. Protocol including ICFs got approval from the Institutional Review Board of Bangladesh Medical Research Council (BMRC/NREC/2022-2025/336) on September 08, 2024. The outcome of this study is to evaluate the effects of telenursing intervention by controlling HbA1c. Investigators set various secondary endpoints including feasibility. By making self-supported decisions, the patients will be able to manage their diet, exercise and medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed as type 2 diabetes
* Both sexes
* Age18-75 years old
* Who will have a smartphone or mobile phone
* Who are willing to participate / give us the consent

Exclusion Criteria:

* Patients who have been diagnosed as Type 1 and gestational diabetes
* Patients whose diabetes is secondary causes
* Patients who have complication of CKD stage 5
* Patients whose HbA1c is less than 7.0% past 1 year with CKD stage 1 or 2, no complications or complications with good control, having enough knowledge (had education before) and implemented good practice regarding diabetes management assessed by the research nurses (hereafter "the nurses")
* Disabled persons who need other person's support for daily living

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | From enrollment to 6 months
  Change HbA1c level between baseline and endline.

SECONDARY OUTCOMES:
Change the self-efficacy | From enrollment to 6 months
  Self-efficacy is measured by the Diabetes Management Self-Efficacy Scale, 5 domain, 20 questions, scale 1-10, higher number indicates more self efficacy
Operational feasibility of the system (Qualitative) | From enrollment to 6 months
  Interview to the nurses, PHC staff Any issues and obstacles
Patient feasibility (qualitative and quantitative) | From enrollment to 6 months
  Engagement rate, Follow-up rate, Satisfaction, Nurse education, Education booklet used, Self-monitoring booklet used, Material will be combined to report patient feasibility. Satisfaction scale has 6 items, 0-5 point, higher point indicates better outcome.
Fasting blood sugar or random blood sugar | From enrollment to 6 months
  Change the value of fasting blood sugar or random blood sugar from baseline to endline
Hospitalized by complication | From enrollment to 6 months
  Count the number of hospitalization
Economical evaluation | At 6th month
  Cost-effectiveness analysis by using questionnaire
Behavior modification (quantitative and qualitative) | From enrollment up to 6 months
  Achievement of monthly set goals, Behavior change (Lifestyle behavior questionnaire), 0-5 score, higher is better
Blood pressure | From enrollment up to 6 months
  Change the value of blood pressure from baseline to endline
Body mass index | From enrollment up to 6 months
  Change the value of body mass index from baseline to endline
Non-high-density lipoprotein cholesterol | From enrollment up to 6 months
  Change the value of non-high-density lipoprotein cholesterol from baseline to endline
Triglyceride | From enrollment up to 6 months
  Change the value of triglyceride from baseline to endline
Estimated glomerular filtration (eGFR) | From enrollment up to 6 months
  Change the value of estimated glomerular filtration (eGFR) from baseline to endline
Urine albumin | From enrollment up to 6 months
  Change the value of urine albumin from baseline to endline
Newly diagnosed diseases (any) | From enrollment up to 6 months
  Count the number of newly diagnosed diseases
Medication/treatment change | From enrollment up to 6 months
  Count the times of medication/treatment change and describe the change (better or worse)
Death | From enrollment up to 6 months
  Count the number of death participants
Adverse events | From enrollment up to 6 months
  Count the number of all adverse events
Compliance of eye check (clinic visit), ECG (cardiovascular check) and Lab test | From enrollment up to 6 months
  Count the number of participants who follow nurses' advice to visit eye check, ECG check and laboratory testing

CONTACTS AND LOCATIONS:
Locations (1):
- Grameen Caledonian College of Nursing (GCCN), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
IPD not be shared to maintain the individual participants privacy.

REFERENCES:
- [Derived] Moriyama M, Huq KATME, Mondol L, Mita AR, Nahar NS. Telenursing Health Education and Lifestyle Modification Among Patients With Diabetes in Bangladesh: Protocol for a Pilot Study With a Quasi-experimental Pre- and Postintervention Design. JMIR Res Protoc. 2025 May 9;14:e71849. doi: 10.2196/71849. PMID 40343747